CLINICAL TRIAL: NCT03649607
Title: Pilot Implementation Trial of Accelerated Resolution Therapy for Treatment of Post-Traumatic Stress in HIV Positive Immigrant, Refugee and Undocumented Africans, Caribbean and Black Canadians
Brief Title: Accelerated Resolution Therapy for HIV Positive African, Caribbean and Black
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18028
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: HIV; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerated Resolution Therapy (Other): Participants will complete a clinical intake assessment before meeting with the therapist and initiating the ART® protocol. Participants will receive the ART intervention over a 21-day period, where imaginal exposure and imagery re-scripting will be used replace previous traumatic experiences. The ART intervention will be assessed through pre- and post-test measures at 60-days post enrolment.
  Interventions: Other: Accelerated Resolution Therapy

INTERVENTIONS:
Other: Accelerated Resolution Therapy — ART was developed to treat both physiological and cognitive aspects of PTSD, which has been described as a consequence of failed memory processing. The use of Voluntary Image Replacement (VIR) parallels imaging re-scripting in which a preexisting negative mental image is transformed into a more benign image. This has been successfully used to treat survivors of traumatic industrial accidents suffering from PTSD. Participants will complete five sessions over a 21-day period.

SUMMARY:
Nearly two-thirds of ACB people living in Ontario are classified as immigrant, refugee or undocumented [non-status/NS] (IRNS) individuals. IRNS people are more likely than the general population to be exposed to events that are associated with posttraumatic stress disorder (PTSD). Furthermore, the diagnosis of HIV is itself a traumatic life event. Nonetheless, significant gaps remain regarding the best strategies for supporting trauma-informed care among ACB IRNS individuals with HIV. Accelerated Resolution Therapy (ARTh) is an exposure-based therapy that incorporates rapid eye movements in a standardized administration over 1-5 sessions. ARTh is an effective brief treatment for PTSD symptoms; but, it's range of therapeutic benefit when applied to people with co-morbid HIV infections is unknown. No studies have leveraged neuroimaging to validate the self-reported empirical therapeutic benefit of ARTh. The investigators propose to investigate the implementation of ARTh, including understanding factors influencing its therapeutic outcomes. The three specific aims of this study are to (1) identify factors influencing the response to ARTh (2) identity neuroimaging indicators for treatment effects of ARTh, and (3) to identify factors influencing ARTh implementation. The investigators will conduct a pre-/post- evaluation of intervention outcomes of ARTh implemented in a sample (n=40) of HIV-positive ACB IRNS ages 18-45 years (Aim 1). The investigators will use statistical analyses to identify factors that may moderate the treatment response of ARTh on PTSD symptoms, HIV symptoms distress and quality of life (Aim 1). The investigators will use diffusion tensor imaging and resting state functional magnetic resonance imaging (fMRI) metrics to assess structural and functional connectivity and examine their associations with PTSD symptoms and HIV symptom distress (Aim 2). Finally, the investigators will use process measures to study two specific implementation factors (acceptability and appropriateness) regarding ARTh use in this population. As a consequence of this research, the investigators expect to generate data that will be used to refine an ARTh implementation protocol that will be integrated into an adaptive implementation trial to reduce gaps in the HIV care continuum through the use of intervention packages for ACB people customized to the individual's needs.

DETAILED DESCRIPTION:
STUDY OVERVIEW - PURPOSE AND BACKGROUND

African, Caribbean and Black (ACB) individuals represent only 4.7% of Ontario's population, yet account for 30% of HIV prevalence in the province. Nearly two-thirds of ACB people living in Ontario are classified as immigrant, refugee or non-status (IRNS) individuals. IRNS people are more likely than the general population to be exposed to events that are associated with posttraumatic stress disorder (PTSD). Furthermore, the diagnosis of HIV is itself a traumatic life event. Nonetheless, significant gaps remain regarding the best strategies for supporting trauma-informed care among ACB IRNS individuals with HIV. For example, IRNS women are more likely than Canadian-born women to have experienced rape, non-sexual physical assault, and civil conflict. ACB IRNS men who have sex with men (MSM) are more likely than non-MSM to have emigrated to Canada as asylum-seekers after fleeing some form of persecution or imminent threat in their countries of origin. Furthermore, while it is known that stigma contributes to exacerbation and severity of HIV symptoms-via the activation of physiological stress responses-there is no known intervention that has been shown to interrupt the pathway by which HIV stigma effects stress and HIV symptoms. Accelerated Resolution Therapy (ART®) is an exposure-based therapy that incorporates rapid eye movements in a standardized administration over 5 sessions in a 3-week period. ART® is effective brief treatment for PTSD symptoms; but, it's range of therapeutic benefit when applied to people with HIV infections is unknown. Although evidence shows that the amygdala is the brain region most reactive to changes in stress stimuli, it remains unknown if therapeutic responses can be reliably validated with biomarkers. No studies have leveraged neuroimaging to validate the self-reported empirical therapeutic benefit of ART®.

The purpose of this study is to investigate the implementation of ART®, including understanding factors influencing its therapeutic outcomes.

The central hypothesis is that ART® will reduce HIV symptom distress by down-modulating the effects of stigma and posttraumatic stress-leading to improved self-reported quality of life. The hypothesis is based on previous research showing that adaptive coping strategies buffer the effects of stigma on stress, as well as evidence from a randomized trial of ART® which demonstrated statistically significant treatment effects for trauma related distress (d=1.88), anxiety (d=1.62), and depression (d=1.41), as well as a clinically meaningful 23-point reduction on the civilian PTSD checklist.[5] The investigators will investigate our central hypothesis by pursuing the following specific aims in a sample of ACB immigrant, refugee and non-status people with HIV.

1. Identify factors influencing the response to ART®
2. Identity neuroimaging indicators for treatment effects of ART®
3. Identify factors influencing ART® implementation

The secondary purpose of this study is to determine if ART® treatment of posttraumatic stress symptoms can decrease inflammation and its effects on HIV symptoms.

ELIGIBILITY:
1. Inclusion Criteria:

   A person will be eligible for study participation if they:
   * identify as Black African, Caribbean and/or Canadian
   * are able to consent to participate/have capacity to consent
   * have previously been diagnosed with HIV
   * score >33 on the PTSD Checklist - Civilian (PCL-5)
   * currently live in the Greater Toronto metropolitan area
   * can speak and understand either English or French
   * are on stable combination antiretroviral therapy for the past six months or more
2. Exclusion Criteria:

A person will be excluded from this study if they meet any of the following conditions:

* born in Canada
* unable to consent to provide documentation of HIV seropositive status
* unable to consent to an MRI, including intolerance due to claustrophobia
* are older than 50 years old.
* have a major psychiatric disorder likely to impede treatment (e.g. psychosis), current suicidal ideation, current treatment for substance addiction, or diagnosis of eye movement disorder.
* severe premorbid or comorbid psychiatric disorders. Among these exclusions are a diagnosis of schizophrenia; bipolar disorder and active depression that will confound the neurological assessments. Subjects with a mild or stable depression including those on stable tricyclic antidepressants, serotonin-reuptake antagonists, or monoamine oxidase (MAO) inhibitors are eligible to enroll.
* chronic seizures, stroke not consistent with cerebral small vessel disease (CSVD), head trauma resulting in loss of consciousness >30 min, and multiple sclerosis.
* brain infection (except for HIV-1), including any fungal meningitis, toxoplasmosis, progressive multifocal leukoencephalopathy. Subjects with any space-occupying brain lesions requiring acute or chronic therapy, for example Central nervous system (CNS) lymphoma, will be excluded from participation.
* metallic implant, e.g., in skull, cardiac devices that do not meet safety standards for MRI

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
HIV Symptom Distress Scale (SDS). | Symptom distress score 60 days post the study start date.
  This 20-item instrument is used to measure overall HIV symptom frequency, distress and clinically relevant clusters. Participants are asked to indicate which of the 20 symptoms they have experienced in the past 2 weeks. Participants are then asked to rate symptom that are present, on the extent to which the symptoms are bothersome (0=do not have symptom; 25=have symptom, but no bother; 50=have symptom, little bother; 75=have symptom, bothers me some; 100= have symptom, bothers me a lot). Scores range from 0 to 100. Higher scores indicate greater symptom distress.

SECONDARY OUTCOMES:
HIV Associated Neurocognitive Disease (HAND). | Composite Z-score 60 days post the study start date.
  The HAND assessment includes a battery of measures commonly used to evaluate neurocognitive functioning in 6 domains: executive function, speed of information processing, attention and working memory, and learning memory. The neurocognitive evaluation will be performed by trained staff and supervised by Dr. Adwoa Agyei with consultation from Dr. Giovanni Schifitto.
  The assessment will include tests of:
  * Executive Function using "Trailmaking Test Part B, Stroop Interference task"
  * Speed of Information Processing using "Symbol Digit Modalities Test and Stroop Color Naming"
  * Attention Memory using "CalCAP(CRT4) and WAIS-III Letter-Number Sequencing"
Working and learning memory | Composite Z-score 60 days post the study start date.
  Patient's learning and working memory will be assessed using the following tests: Rey Complex Figure Test Immediate Recall, Rey Auditory Verbal Learning, Test RAVLT Delayed Recall, Rey Complex Figure Test Delayed Recall.
  The working and memory test will be part of the HAND assessment.

OTHER OUTCOMES:
HIV Viral Load | Number of viral particles per ml of plasma 60 days post the study start date.
  The investigators will assess the volume of HIV in serum measured using reverse transcriptase polymerase chain reaction (RT PCR). The HIV viral load is a measure of the number of viral particles per ml of plasma. Higher numbers of HIV viral copies indicate inadequate viral suppression and insufficient immune function. The data will be entered directly into REDCap by the St. Michael's Hospital lab personnel. The investigators will code viral suppression as <50 HIV copies/mL of blood as "=yes" and ≥50 "=no."
Post Traumatic Stress Disorder (PTSD) Checklist - Civilian Version (PCL-5) | Posttraumatic stress score 60 days post the study start date.
  This 20-item measure assesses symptoms of posttraumatic stress. It assesses an individual's symptoms based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for PTSD. The PCL-5 focuses on four aspects of distressing memories: re-experiencing the event, avoidance, mitigation and hyperarousal. The scale uses a 5-point Likert scale that ranges from 0 to 4 (0 [Not at all]; 1[A little bit]; 2 [Moderately]; 3 [Quite a bit]; 4 [Extremely]) to rate each of the 20 items on the degree to which symptoms were present and bothersome in the prior 30-days. For PTSD diagnosis, the score must be above certain cut-point indicating moderate to high symptom severity. The PCL-5 showed good internal consistency in a study with HIV-positive patients in Ghana (α=0.79).
HIV/AIDS Related Quality of Life | Quality of life measure 60 days post the study start date.
  There is a 34-item tool that measures experiences in overall function, life satisfaction, health and financial worries, worries about medication, HIV disclosure, living with HIV and doctor satisfaction in the past month. Check boxes to 5 specific answers (All the time; A lot of the time; Some of the time; A little of the time; None of the time) are used to measure and evaluate quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: LaRon Nelson, PhD, RN, FNP, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No
No one outside of the principal investigator, research assistant, therapists administering ART®, study medical director and a medical provider with a clinical "need to know" will have access to any identifiable data. The research assistant will need access to basic identifying data such as name, phone number for follow-up contact purposes to aid in recruitment, enrollment and data collection. If an urgent clinical issue arises (such as, a participant experiencing acute psychological distress) it may be necessary to link the participant's contact information to subject's identity in order to provide clinical follow-up. No data will be shared without the participant's written informed consent to release medical information. It is in keeping with the principle of beneficence to ensure continuity of care by making it possible (not mandatory) for participants to share information with the medical provider.